CLINICAL TRIAL: NCT00993408
Title: A Multi-centre, Multinational, Open-label, Single-dose Acute Hemodynamic Study Followed by Multi-centre, Multinational, Randomized, Double-blind, Parallel-group, Placebo Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy (Proof-of-concept) of ACT-293987 (NS-304) in the Treatment of Pulmonary Arterial Hypertension in Subjects Aged 18 Years and Over
Brief Title: Study of ACT-293987 (NS-304) in Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: NS-304/-02
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACT-293987 (NS-304) and matching placebo (Experimental): Subjects will be randomized to the study following screening.
  Each subject will then undergo an acute hemodynamic study with right heart catheterization after a single oral administration of ACT-293987 (NS-304)on Day 0. The objectives are to collect data about the drug effect on the right heart hemodynamic parameters (PVR, calculated SVR and PVR/SVR) measured by right heart catheterization after single oral dose administration of NS-304 and to assess the safety and tolerability of a single oral dose of NS-304.
  Interventions: Device: ACT-293987 (NS-304)

INTERVENTIONS:
Device: ACT-293987 (NS-304)

SUMMARY:
This is a multi-centre, multinational, open-label, single-dose acute hemodynamic study followed by randomized, double-blind, parallel-group, placebo controlled study. Eligible subjects will undergo an open-label, single-dose acute hemodynamic study with ACT-293987(NS-304) and 21 weeks of double-blind treatment during which subjects will receive either ACT-293987 (NS-304) or placebo b.i.d. Subjects who have completed the double-blind study can enter the open extension study (separate protocol) and receive administration of ACT-293987 (NS-304) if the subject wishes and the Investigator considers it appropriate.

DETAILED DESCRIPTION:
This is a multi-centre, multinational, open-label, single-dose acute hemodynamic study followed by a randomized, double-blind, parallel-group, placebo controlled study. Eligible subjects will undergo screening followed by randomized allocation to treatment group for the double-blind study, followed in turn by immediate enrollment in an open-label, single-dose acute hemodynamic study with ACT-293987 (NS-304) and 21 weeks of double-blind treatment during which subjects will receive either ACT-293987 (NS-304)or placebo twice daily (b.i.d.). Subjects who have completed the double-blind study can enter the open extension study and receive administration of ACT-293987 (NS-304) (separate protocol)if the subject wishes and the investigator considers it appropriate.

Unblinding will occur on a subject-by-subject basis when the Week 17 data for the subject have been fixed.

Approximately 44 subjects are to be randomized in a ratio of 3:1 to the two treatment groups, ACT-293987 (NS-304) and placebo (33 subjects to ACT-293987 (NS-304) and 11 subjects to placebo).

Subjects will be randomized to the study following screening.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age or older with symptomatic PAH despite treatment with anticoagulants, calcium channel blockers, diuretics, cardiac glycosides, supplemental oxygen, endothelin-receptor antagonists and/or phosphodiesterase inhibitors. Endothelin receptor antagonists and phosphodiesterase inhibitors must have been used at a stable dose for more than 12 weeks before screening.
2. Subjects with idiopathic PAH, familial pulmonary arterial hypertension and PAH associated with collagen vascular disease, corrected congenital vitium (congenital systemic to pulmonary shunts surgically repaired at least five years before) or anorexigen use.
3. Diagnosis of PAH established according to the standard criteria:

   1. Resting mean pulmonary arterial pressure > 25 mmHg.
   2. PVR > 240 dynes s/cm5.
   3. Pulmonary capillary wedge pressure or left ventricular end diastolic pressure < 15 mmHg.
4. PVR > 400 dynes s/cm5.
5. Two 6MWTs between 150 and 500 m (inclusive) with the variation in 6MWT within ± 15% between the two tests despite other treatments for PAH.

   - Two 6MWT values are needed. Only one 6MWT should be performed at screening for confirmation of eligibility if 6MWT has been previously conducted within six weeks of the screening visit unless the subject was taking another investigational drug or participating in a specific training and exercise programme at the time of the previous test.
6. Subjects who are able and willing to refrain from sunbathing, prolonged sun exposure, and solarium use, and to limit skin and eye exposure to sunlight using appropriate precautions (protective clothing, sunscreen and sunglasses) from the first dose until 14 days after study drug discontinuation.

Exclusion Criteria:

Subjects will not be entered in the study for any of the following reasons:

1. Subjects with clinically unstable right heart failure within the last three months (NYHA Class IV).
2. Subjects who have received or have been scheduled to receive long-term treatment with epoprostenol within three months before screening.
3. Hypotensive subjects (systemic systolic blood pressure < 85 mmHg).
4. Subjects with PAH associated with portal hypertension, Human Immunodeficiency Virus infection or unrepaired congenital systemic to pulmonary shunts.
5. Subjects with ventilation-perfusion lung scan or pulmonary angiography indicative of thromboembolic disease.
6. Subjects with significant obstructive (forced expiratory volume in one second [FEV1]/forced vital capacity [FVC] < 70% predicted) or restrictive (total lung capacity < 70% predicted) lung disease.
7. In collagen vascular diseases, subjects with significant interstitial disease (FVC < 70% predicted).
8. Subjects with evidence of left sided heart disease.
9. Subjects with moderate or severe hepatic impairment (Child-Pugh B and C).
10. Subjects with clinically significant chronic renal insufficiency (estimated creatinine clearance < 30 mL/minute, or serum creatinine > 2.5 mg/dL).
11. Subjects who are receiving or have been receiving any investigational drugs within 30 days before screening.
12. Subjects with musculoskeletal disorder limiting ambulation.
13. Females who are breast-feeding, pregnant or plan to become pregnant during the study and females who are not using a highly effective method of birth control (failure rate less than 1% per year) such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomised partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-04-30 (Actual); Primary Completion 2009-06-30 (Actual); Study Completion 2009-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of hemodynamic parameters after single oral dose of ACT-293987. | 17 weeks
Proof-of-concept assessment of the efficacy of ACT-293987 in subjects with PAH by measuring the change from baseline in the PVR at Week 17 compared to placebo. | 17 weeks

SECONDARY OUTCOMES:
Safety and tolerability of a single oral dose of ACT-293987. | 17 weeks
Assessments of preliminary efficacy of ACT-293987 regarding 6 minute walk test (6MWT), proportion of subjects with aggravation of PAH, hemodynamic parameters other than PVR | 17 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- Medizinische Universitat Wien, Universitatsklinik fur Innere Medizin II, Kardiologie, Vienna, Austria
- Gasthuisberg University Hospital, Pneumology, Leuven, Belgium
- Hopital Antoine Beclere, Pneumologie, Paris, France
- Department of Respiratory Medicine, Hannover Medical School, Hanover, Germany
- Semmelweis University, Clinic of Pulmonology, Budapest, Hungary
- Hospital Sant'Orsola Malpighi, Cardiology's Department, Bologna, Italy
- Instytut Gruzilcy i Chorob Pluc, Klinika Chorob Wewnetrznych Klatki Piersiowej, Warsaw, Poland
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Derived] Simonneau G, Torbicki A, Hoeper MM, Delcroix M, Karlocai K, Galie N, Degano B, Bonderman D, Kurzyna M, Efficace M, Giorgino R, Lang IM. Selexipag: an oral, selective prostacyclin receptor agonist for the treatment of pulmonary arterial hypertension. Eur Respir J. 2012 Oct;40(4):874-80. doi: 10.1183/09031936.00137511. Epub 2012 Feb 23. PMID 22362844